CLINICAL TRIAL: NCT05310799
Title: Treating Children With Arthritis According to Their Individual Probability of Outcomes and Response to Treatments
Brief Title: Personalized Estimates of Response and Severity Outcomes in Newly-diagnosed JIA
Acronym: PERSON-JIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Lori Tucker, Head, Pediatric Rheumatology, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-00593
Record Dates: First submitted 2021-11-29; First posted 2022-04-05 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; Arthritis, Juvenile; Arthritis; Shared decision making; Clinical outcomes; Canada; PERSON-JIA; PERSON JIA
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Best Practice (No Intervention): Physicians randomized to this arm will provide current care and treatment decisions with patients will be made in accordance with current best practices. Will not engage in structured shared decision making (SDM) discussion and will not have access to PERSON-JIA Reports.
  Patients will be consented to enroll in the CAPRI Registry at the clinic visit when they are diagnosed. Registry enrollment will allow collection and input of clinical data into the Registry.
  Clinic visit and discussion will remain unchanged for physicians, patients and their families. Questionnaires will be collected at enrollment, at the second visit and a 6-month and 12-month follow-up visits.
- Shared Decision Making (SDM) (Experimental): Physicians will use the PERSON-JIA Report to guide discussions with the newly diagnosed patient and family. The intervention will not dictate the use of specific medications or treatment strategies, only facilitate better informed treatment choices according to patient circumstances.
  The intervention is a structured SDM discussion between physician and family, occurring at the time of the child's JIA diagnosis. Discussion is guided by the PERSON-JIA Report, which is generated in real time, on the physician's smart phone.
  Patients newly-diagnosed with JIA will be consented to both enrollment in the CAPRI Registry and enrollment in the PERSON-JIA trial.
  Clinic visit and discussion between the physician, patient and family will be facilitated by the PERSON-JIA report to support a shared decision making process. Questionnaires will be collected at enrollment, at the second visit and at 6-month and 12-month follow-up visits.
  Interventions: Other: Shared Decision Making (SDM)

INTERVENTIONS:
Other: Shared Decision Making (SDM) — The intervention is a structured SDM discussion between physician and family, occurring at the time of the child's JIA diagnosis and clinic visit. Discussion will be guided by a discussion guide and the PERSON-JIA Report, which is generated in real time on the physician's smart phone.
  Arms: Shared Decision Making (SDM)

SUMMARY:
The PERSON-JIA Trial is a cluster-randomized trial testing the use of Shared Decision Making (SDM) with families for treatment of children with arthritis. The intervention is a discussion between physicians and families at the time of diagnosis that uses computer-generated personalized outcome reports generated by previously developed prediction algorithms.

By using information provided by thousands of families, the investigators have developed a way of providing answers to common questions asked by patients and their families at diagnosis.

We will test whether a structured discussion and shared decision between families and doctors (guided by the patient's personal report) will improve the tailoring of treatment to the child and control of their disease. The personal report is called the PERSON-JIA report and presents the child's expected disease severity, the likelihood the child will be arthritis free by age 18 and the chance treatments will be effective and/or have side effects. This way, answers to these questions can be shared by physicians and families to weigh potential benefits and harms according to family values and preferences.

The investigators expect that using the personalized report in a frank and thoughtful discussion will help physicians and families make better decisions about managing the child's disease. This in turn will result in better disease control, greater family engagement and satisfaction with care and better-tailored treatment. If so, this will be a ground-breaking way of using information provided by families and doctors to improve the care provided to and the outcomes of children with arthritis in Canada.

DETAILED DESCRIPTION:
The PERSON-JIA (Personalized Estimates of Response and Severity Outcomes in Newly-diagnosed Juvenile Idiopathic Arthritis) trial, will test an innovative shared decision making (SDM) intervention - a structured discussion, between physician and family, of the likely outcomes/response to treatments, as predicted by Personalized Prediction Algorithms (PPA), presented in a graphical summary.

Juvenile Idiopathic Arthritis (JIA) is chronic arthritis of unknown cause starting before the 16th birthday. At present, evidence does not suggest that any single treatment approach for treating JIA is clearly superior, and current practice guidelines recommend Shared Decision Making (SDM) with families to select treatment. SDM requires a realistic appreciation of disease severity along with the likely benefits vs. harms associated with treatment options, and to then weigh these factors according to the family's values and preferences.

To facilitate SDM, the investigators have built and validated PPA using data from previous Canadian JIA cohorts. As compared to treatment algorithms/flowcharts that tell physicians what to do, PPA are mathematical models that calculate the probability of outcomes for a child, based on their clinical presentation.

The investigators have also established a Canadian Alliance of Pediatric Rheumatology Investigators (CAPRI) JIA Registry, which supports point of care data entry using smartphones/tablets. After data is entered in the registry for a newly diagnosed patient, PPA produce a graphical report depicting that child's probability of severe disease, remission in adulthood, and response and side effects with different treatments. This randomized controlled trial (RCT) will test the impact on JIA outcome of a SDM intervention that uses this graphical report to better tailor treatment to the child and family.

The investigators hypothesize that compared to current standard care, use of this SDM intervention will lead to improved JIA disease control at 6 months via increased family engagement, greater satisfaction with treatment decisions, optimal tailoring of treatment to the child, and consistent adherence to the treatment plan.

PERSON-JIA is a registry-based, pragmatic, cluster-randomized (by physician) adaptive trial.

Pediatric rheumatologists from all pediatric rheumatology sites in Canada who agree to participate will be matched with another rheumatologist (by practice size, province and years in practice). There will be a one to one randomization of physicians to the intervention group or control group.

Patients will be placed into the intervention or control group dependent on which group their pediatric rheumatologist has been randomized to. Control pediatric rheumatologists will practice standard care without the PPA or shared decision making discussion, but will still enroll all their new JIA patients into the CAPRI JIA Registry.

Pediatric rheumatologists in the intervention group will have structured SDM discussions with the patient and family using the graphical PERSON-JIA report generated by PPA, at the time of diagnosis. The intervention will occur once, at the time of initial treatment decision making. Patients in the intervention arm of the study may have slightly longer clinic visits to account for a tailored, shared decision making discussion regarding their disease course and treatment options.

The primary outcome will be inactive or minimally active disease 6 months after enrolment, defined using the clinical Juvenile Arthritis Disease Activity Score 10 (cJADAS10). CJADAS10 scores go from 0=best to 30=worst. Inactive or minimally active disease is 2.5 or less for patients with >4 joints involved and 1.5 or less for patients with 1-4 joints.

Secondary outcomes include inactive or minimally active disease 12 months after enrolment; quality of life and function; implementation of treatment plan; parent and doctor assessments of how much decisions were shared; parent's knowledge, value alignment, uncertainty and satisfaction with the decision; and intervention fidelity (analysis of medical encounter audio recordings).

The primary statistic will be the odds ratio of patients achieving inactive or minimally active disease at 6mos, adjusted for clustering effects and baseline cJADAS10 scores.

ELIGIBILITY:
Physicians (Inclusion):

1. Licensed to practice pediatric rheumatology in Canada;
2. Providing care for children with JIA at least once a month;
3. Consent to be randomized and to implement the SDM intervention for the duration of the trial, if randomized to the intervention arm;
4. Commit to propose enrollment in the Registry to all their newly diagnosed patients with JIA during the trial.

Physicians (Exclusion):

1. Fellows-in-training;
2. Physicians planning to retire within 2 years.

Patient (Inclusion):

1. Consent to include their information in the CAPRI JIA Registry;
2. Consent to the PERSON-JIA trial and answering additional questionnaires to assess decision making;
3. Allow recording of their medical encounter (if selected at random);
4. JIA fulfilling International League of Associations for Rheumatology (ILAR) criteria;
5. Newly diagnosed (within the last month);
6. Diagnosed by a pediatric rheumatologist participating in the PERSON-JIA study;
7. Not yet receiving treatment, or received only Non-Steroidal Anti-Inflammatory Drugs (NSAIDS) or joint injections;

Patient (Exclusion):

1. Systemic arthritis category of JIA (it requires a different treatment approach);
2. Family is unable to complete study forms in English or French;
3. Patients who have already started systemic corticosteroid or any Disease Modifying Anti-Rheumatic Drug (DMARD).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 842 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with Inactive or Minimally Active Disease at 6 months. | 6 months after enrollment
  Proportion of patients attaining inactive or minimally active disease within 6 months of study enrollment, defined as a cJADAS (Clinical Juvenile Arthritis Disease Activity Score 10) of 2.5 or less for patients with >4 joints involved and 1.5 or less for patients with 1-4 joints involved.
  The cJADAS10 is the sum of the number of active joints (to a maximum of 10), the Physician Assessment of Disease Activity (PGADA 0 to 10), and the Parent Global Assessment of well-being (0-10).

SECONDARY OUTCOMES:
Proportion of children with Inactive or Minimally Active Disease at 12 months. | 12 months after enrollment
  Proportion of patients attaining inactive or minimally active disease within 12 months of study enrollment, defined as a cJADAS (Clinical Juvenile Arthritis Disease Activity Score 10) of 2.5 or less for patients with >4 joints involved and 1.5 or less for patients with 1-4 joints involved.
  The cJADAS10 is the sum of the number of active joints (to a maximum of 10), the Physician Assessment of Disease Activity (PGADA 0 to 10), and the Parent Global Assessment of well-being (0-10).
  The comparison at 6 months and at 12 months will be done using a mixed-effects logistic regression model that accounts for the clustering of patients by physician, the paired randomization to intervention or control, the JIA category and the three cJADAS10 components.
Change in Parent-Reported Health-Related Quality of Life | From enrollment to 6 and 12 months
  Mean change in parent-reported health-related quality of life (QoL), assessed according to the Juvenile Arthritis Quality of Life Questionnaire (JAQQ). JAQQ scores go from 1=best to 7=worst.
Change in Patient-Reported Health-Related Quality of Life | From enrollment to 6 and 12 months
  Mean change in patient-reported health-related quality of life (QoL), assessed according to the Quality of my Life Scale, unless parents state the patient is too young to answer the questionnaire. Scores go from 0=worst to 10=best.
Change in cJADAS10 score | From enrollment to 6 and 12 months
  Mean change on the clinical Juvenile Arthritis Disease Activity Score with 10 joints (cJADAS10) and its components. Scores go from 0=best 30=worst.
Change in functional impairment | From enrollment to 6 and 12 months
  Mean change in functional impairment, assessed according to the Childhood Health Assessment Questionnaire Disability Index (CHAQ). Scores go from 0= no disability to 3.0= severe disability.
Change in Health Utilities | From enrollment to 6 and 12 months
  Mean change in health utilities, assessed according to the European Quality of Life 5 Dimension Scale for Youth (EQ-5D-Y). Score goes from 0=dead to 1.0=perfect health
Parent assessment of decision making | 1-3 months
  Parents assessment of how much decision were shared according to the 9-item Shared Decision Making Questionnaire (SDM-Q9). Scores go from 0=no shared decision making to 100=maximal sharing of decisions.
Parent assessment of decisional conflict | 1-3 months
  Parent's decision-related knowledge, value-alignment, uncertainty and satisfaction, measured with the Decisional Conflict Scale (DCS) at Visit 2. From 0= no decisional conflict to 100=maximum decisional conflict.
Doctor assessment of decision making | 1-3 months
  Physicians will answer the physician version the 9-item Shared Decision Making Questionnaire (SDM-Q-DOC), at the first follow-up visit after patient enrollment (Visit 2). Scores go from 0=no shared decision making to 100=maximal sharing of decisions.
Proportion of children receiving recommended treatment | 1-3 months
  The proportion of children receiving the recommended treatment by visit 2. The treatment plans are noted in the Registry at Visit 1 as 'Changes Recommended Today.' Listed medications will be compared to the medications the patient is actually taking at Visit 2. If the lists coincide, the patient will be counted as treatment implemented.
Intervention Fidelity | The first patient enrolled and another selected at random within the next 24 weeks
  Fidelity of the intervention will be assessed by thematic analysis of a sample of audio recordings of medical encounters, and the Observing Patient Involvement (OPTION) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lori B Tucker, MD, Principal Investigator — University of British Columbia Department of Pediatrics
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada